CLINICAL TRIAL: NCT07315555
Title: Efficacy of Oral Nigella Sativa as Adjuvant Therapy in Children With Moderate Persistent Asthma
Acronym: Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Zaki Elmeazawy, Associate professor of pediatrics, Tanta University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR131072/11/25
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Community Acquired Pneumonia
Keywords: Nigella sativa; Pneumonia; Pediatric
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Nigella sativa oil; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard asthma Controller Therapy Only (Active Comparator): 30 children with moderate persistent asthma receiving standard controller therapy consisting of a combined low-dose inhaled corticosteroid (ICS) and long-acting β2-agonist (LABA), administered by metered-dose inhaler with spacer.
  Interventions: Dietary Supplement: Nigella sativa Oil Capsules (100 mg/kg/day); Dietary Supplement: Nigella sativa Oil Capsules (50 mg/kg/day)
- Standard Therapy + Nigella sativa (50 mg/kg/day) (Experimental): 30 children with moderate persistent asthma receiving standard controller therapy plus Nigella sativa oil capsules at a dose of 50 mg/kg/day as adjunct therapy.
  Interventions: Dietary Supplement: Nigella sativa Oil Capsules (100 mg/kg/day); Drug: Fluticasone / Long-Acting Beta-2 Agonist Combination
- Standard Therapy + Nigella sativa (100 mg/kg/day) (Experimental): 30 children with moderate persistent asthma receiving standard controller therapy plus Nigella sativa oil capsules at a dose of 100 mg/kg/day as adjunct therapy.
  Interventions: Dietary Supplement: Nigella sativa Oil Capsules (50 mg/kg/day); Drug: Fluticasone / Long-Acting Beta-2 Agonist Combination

INTERVENTIONS:
Dietary Supplement: Nigella sativa Oil Capsules (100 mg/kg/day) — Nigella sativa oil administered orally in capsule form at a dose of 100 mg/kg/day as adjunct therapy.
  Arms: Standard Therapy + Nigella sativa (50 mg/kg/day); Standard asthma Controller Therapy Only
Dietary Supplement: Nigella sativa Oil Capsules (50 mg/kg/day) — Nigella sativa oil administered orally in capsule form at a dose of 50 mg/kg/day as adjunct therapy.
  Arms: Standard Therapy + Nigella sativa (100 mg/kg/day); Standard asthma Controller Therapy Only
Drug: Fluticasone / Long-Acting Beta-2 Agonist Combination — Low-dose inhaled corticosteroid (fluticasone propionate 200 µg/day) combined with a long-acting beta-2 agonist (two puffs every 12 hours), administered via metered-dose inhaler with spacer.
  Arms: Standard Therapy + Nigella sativa (100 mg/kg/day); Standard Therapy + Nigella sativa (50 mg/kg/day)

SUMMARY:
Complementary and adjunctive therapies are increasingly being explored to enhance asthma control and reduce airway inflammation. Nigella sativa (black seed) is a medicinal plant used traditionally in multiple regions and has demonstrated anti-inflammatory, immunomodulatory, and bronchodilator effects. Its potential as an adjuvant therapy in asthma has attracted attention in both preclinical and clinical research

DETAILED DESCRIPTION:
We hypothesize that supplementation with Nigella sativa will lead to improved asthma control scores and enhanced pulmonary function parameters in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-18 years
2. Diagnosed with moderate persistent asthma according to the Global Initiative for Asthma (GINA) 2022 guidelines
3. Receiving stable standard controller therapy (inhaled corticosteroids ± long-acting β2-agonists) for at least 4 weeks prior to enrollment
4. Able to perform reproducible spirometry

Exclusion Criteria:

1. History of severe asthma exacerbation requiring ICU admission in the past 3 months
2. Use of systemic corticosteroids within 4 weeks prior to enrollment
3. Known hypersensitivity to Nigella sativa or its components
4. Other chronic respiratory diseases (e.g., cystic fibrosis, bronchiectasis)
5. Significant comorbidities (e.g., cardiac, renal, or hepatic disorders)
6. Inability to comply with study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | 12 weeks
Forced Expiratory Volume in 1 second (FEV₁) | 12 weeks
  Pulmonary function will be assessed using standard spirometry performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines.
Forced Vital Capacity (FVC) | 12 weeks
  Pulmonary function will be assessed using standard spirometry performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines.
FEV₁/FVC ratio | 12 weeks
  Pulmonary function will be assessed using standard spirometry performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines.
Peak Expiratory Flow (PEF) | 12 weeks
  Pulmonary function will be assessed using standard spirometry performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines.

IPD SHARING:
Plan to Share IPD: No